CLINICAL TRIAL: NCT00493441
Title: A Phase II Study of AVN944 in Combination With Gemcitabine for the Treatment of Pancreatic Cancer
Brief Title: AVN944 in Combination With Gemcitabine for the Treatment of Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVN944-006
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — AVN 944

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: AVN944

INTERVENTIONS:
Drug: AVN944 — 150, 200, 250, 300, or 400 mg q12h

SUMMARY:
The study was designed to find the optimum AVN944 dose to use in combination with gemcitabine in patients with pancreatic cancer and see if the combination of the 2 drugs was more effective for treating pancreatic cancer than using gemcitabine alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed adenocarcinoma of the pancreas not eligible for curative intent resection with or without adjuvant radiation therapy
* Measurable disease as defined by RECIST criteria
* No prior chemotherapy for pancreatic cancer including no prior "radiosensitizing" chemotherapy
* Patients are candidates to receive gemcitabine as first line treatment for adenocarcinoma of the pancreas
* Age > 18 years
* Karnofsky Performance Score of less than or equal to 60
* Patients must be recovered from the clinically significant effects of any prior surgery or prior radiotherapy
* Adequate bone marrow, hepatic and renal function as evidenced by:

  * Serum total bilirubin < 2.0 mg/dL
  * AST/ALT (SGOT/SGPT) < 4X the ULN for the reference lab;
  * Serum creatinine < 2.0 mg/dL;
  * ANC > 1.5 x 109/L;
  * Platelet count > 100 x 109/L,
  * Hgb > 9.0 g/dL
* Female patients of childbearing potential as well as fertile men and their partners who agree to use an effective form of contraception during the study and for 90 days following the last dose of study medication (an effective form of contraception is an oral contraceptive or a double barrier method)
* Patients or their legal representatives must be able to read, understand and provide written informed consent to participate in the trial.

Exclusion Criteria:

* Patients with a life expectancy < 3 months
* Patients with known CNS metastases
* Patients with an uncontrolled active infection
* Prior treatment with an IMPDH-inhibitor
* Patients with known hypersensitivity to any of the components of AVN944 or gemcitabine
* History of prior malignancy within the past 5 years except for curatively treated non-melanoma skin cancers; cervical intraepithelial neoplasia, or localized prostate cancer with a current PSA of < 1.0 mg/dL
* Patients who are receiving concurrent investigational therapy or who have received investigational therapy within 14 days of the first scheduled day of dosing (investigational therapy is defined as treatment for which there is currently no regulatory authority approved indication). Clinically significant toxicities from this therapy must have resolved to < Grade 2.
* Patients who are pregnant or lactating
* Myocardial Infarction within the past 6 months
* Patients with clinically significant intraventricular conduction delays
* Any other intercurrent medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* History of solid organ transplant
* Known HIV or Hepatitis B or C (active, previously treated or both)
* Previous treatment under this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Safety | 4 weeks
Pharmacokinetics | Days 1, 8, 15, and 22

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - University of Florida - Shands Cancer Center, Gainesville, Florida
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Joliet Oncology and Hematology Associates, Joliet, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University, New York, New York
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - Chattanooga Oncology and Hematology Associates, Chattanooga, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Sarah Cannon Research Institute -Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer institute, Richmond, Virginia